CLINICAL TRIAL: NCT06301412
Title: Combination of Targeted Temperature Management and Thrombectomy After Acute Ischemic Stroke (COTTIS-2) - a Randomised Controlled Study
Brief Title: Combination of Hypothermia and Thrombectomy in Acute Stroke
Acronym: COTTIS-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Freiburg (Other)
Collaborators: European Union (Other); E+E CRO consulting, Vienna, Austria (Unknown); Center for Medical data science, University of Vienna, Austria (Unknown)
Responsible Party: Principal Investigator, Juergen Bardutzky, Prof. Dr. med. Juergen Bardutzky, University of Freiburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COTTIS-2_Version4.0-13Nov23
Record Dates: First submitted 2024-02-22; First posted 2024-03-08 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Ischemic Stroke; Large Vessel Occlusion; Endovascular Treatment
Keywords: hypothermia; neuroprotection
MeSH Terms: conditions — Ischemic Stroke; Hypothermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVT group (No Intervention): standard endovascular treatment (EVT) for large vessel occlusion (LVO) without hypothermia
- EVT group plus hypothermia group (Active Comparator): standard endovascular treatment (EVT) for large vessel occlusion (LVO) combined with hypothermia
  Interventions: Device: hypothermia

INTERVENTIONS:
Device: hypothermia — hypothermia is started after intubation for endovascular treatment and induced by transnasal cooling (RhinoChill) to a target temperature of 35°C and hypothermia is then maintained at 35°C for 6 hours after recanalisation by surface cooling followed by slow rewarming by 0.2°C per hour to 36.5°C
  Arms: EVT group plus hypothermia group

SUMMARY:
The goal of this clinical trial is to test the combination of hypothermia and endovascular treatment in acute stroke patients with large vessel occlusion.

The main question it aims to answer is: does an additional cooling to 35°C result in a benefit on clinical outcome ? Participants receive immediate cooling using a noninvasive transnasal cooling technique (RhonoChill) and are maintained at 35°C for 6 hours after reopening of the vessel using surface cooling, and then slowly rewarmed.

Researchers will compare the intervention group (hypothermia and endovascular treatment and best medical treatment including iv thrombolysis) and control group (only endovascular treatment and best medical treatment including iv thrombolysis) to see if additional hypothermia leads to a better outcome after 3 months without relevant complications.

DETAILED DESCRIPTION:
Despite the well-established benefit of endovascular treatment (EVT) for acute ischemic stroke due to large vessel occlusion (LVO), more than half of patients treated with EVT remain functionally dependent despite high reperfusion rates. Thus, new strategies such as additional neuroprotection using hypothermia need to be explored, first to bridge time to reperfusion and second, to attenuate reperfusion injury.

Although therapeutic hypothermia has consistently demonstrated robust neuroprotection in animal ischemic-reperfusion models, randomized trials in acute stroke patients have failed to demonstrate the efficacy of induced hypothermia. The reasons for this treatment failure are diverse and include treatment delay, the unfeasibility of inducing and maintaining hypothermia due to intolerance and shivering in awake patients, the missing recanalization in a large proportion of patients, the heterogeneity of patients included, and too deep (32-34°C) hypothermia associated with an increase in side effects.

In the pilot study COTTIS-1, we could demonstrate the feasibility and safety of immediately induced intraischemic hypothermia to 35°C with non-invasive transnasal cooling by RhinoChill® (BrainCool) followed by surface cooling for 6h after recanalization in sedated and intubated patients with LVO undergoing EVT. By combining this cooling technique with thrombectomy we have tried to address the above mentioned reasons for hypothermia failure. In COTTIS-1, the target temperature of 35°C was reached within 30 min, corresponding to a cooling rate of 2.6°C/h. All patients reached the target temperature, and 86% of the patients had reached ≤35°C at recanalization by thrombectomy. 68% of patients had a good outcome (independency) after 3 months. There were only asymptomatic side effects during hypothermia.

As a consequence, the present COTTIS-2 study is planned to evaluate the efficiency of this cooling protocol in a multicentric, randomized, controlled, end-point-blinded study in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Pre-stroke modified Rankin Scale (mRS) 0-2 [7-point scale rating from 0 (no symptoms) to 6 (dead)]
* Acute ischemic stroke with NIHSS >5
* Intracranial occlusion of the M1 or M2 segment of the middle cerebral artery (MCA) or internal carotid artery (ICA) or tandem occlusion on CT-angiography or MR-angiography with indication for endovascular treatment:
* Time window 0-24h:

  1. Last seen normal to groin puncture < 6h: native CT or MRI-DWI with ASPECTS >5
  2. Last seen normal to groin puncture 6-24h or unknown time window: significant mismatch imaging according to the eligibility criteria of the DEFUSE-3 trial

     * Infarct core <70ml (DWI oder CBF<30%)
     * Penumbra > 15ml (Tmax >6sec)
     * Ratio penumbra/core >1.8
* with or without iv thrombolysis with rtPA

Exclusion Criteria:

* Patients with an intranasal obstruction that prevents complete insertion of the nasal cannula should not be treated with the RhinoChill system.
* Known severe hemorrhagic diathesis (International Normalized Ratio (INR) >3.0, partial thromboplastin time (PTT) > 70s, platelet count < 50.000/μl)
* Brain trauma or neurovascular surgery/intervention <3 months
* Severe infection
* Pregnant women or women of childbearing potential (women of childbearing potential with negative pregnancy test may be included)
* Known cerebral vasculitis
* Proof of bleeding in cerebral CT or MRI (cerebral microbleeds in MRI [hypertensive or in the context of cerebral amyloid angiopathy] is permitted).
* Known life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-07-07 (Actual); Primary Completion 2026-03-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
functional outcome | 3 months
  The presence of patients with good neurological outcome after 3 months as defined by modified Rankin Scale (mRS; on which scores range from 0 to 6, with 0 means no symptoms and 6 means death) of 0-2 or back to baseline before stroke

SECONDARY OUTCOMES:
infarction volume | 24 hours
  Infarction volume assessed in the standard CT 24 hours after thrombectomy
increase in infarction | 24 hours
  increase of the infarct core based on imaging at the time of admission (DWI-MRI or CBF<30% of contralateral side at CT-Perfusion) and CT after 24 hours
recanalization result | after thrombectomy and 24 hours
  Recanalization result (by mTICI score: successful recanalization mTICI 2b-3) after thrombectomy (based on angiography during/after thrombectomy) and 24 hours after thrombectomy (based on ultrasound of the cerebral vessels)
neurological improvement | 48 hours
  Change of at least 8 points on the National Institutes of Health Stroke Scale (NIHSS; on which scores range from 0 to 42, with higher scores indicating a greater deficit) at 48 hours after thrombectomy
outcome at discharge | up to 3 months
  modified Rankin Score (mRS; on which scores range from 0 to 6, with 0 means no symptoms and 6 means death) upon discharge/transfer in rehabilitation
shift in functional outcome | 3 months
  ordinal shift across the range of modified Rankin Score (mRS; on which scores range from 0 to 6, with 0 means no symptoms and 6 means death)
very good clinical outcome | 3 months
  Presence of patients with very good clinical outcome after 3 months (mRS 0-1)
mortality | 3 months
  Mortality during acute hospitalisation and after 3 months
Length of ventilation | 3 months
  Length of mechanical ventilation
Length of stay | 3 months
  Length of ICU stay and hospital stay
body temperature | 24 hours
  Temperature at admission, at recanalization, and first 6 hours after recanalization, and at 24 hours
time to groin puncture | baseline, pre-intervention
  Time from arrival until groin puncture
time to recanalization | periprocedurally
  Time from arrival until recanalization

OTHER OUTCOMES:
Occurrence of intracerebral haemorrhage (ICH) | 24 hours
  * Any ICH (subarachnoid, intraparenchymal, intraventricular) on the CT after 24 hours
  * Symptomatic ICH (defined according to SITS-MOST criteria):
  Hematoma >30% of initial infarction volume associated with a clinical deterioration in NIHSS score of at least 4 points within 24 hours after thrombectomy
Complications associated with hypothermia | 24hours
  * Nosebleed and pailing of the nose
  * Periorbital emphysema
  * Pneumocephalus (in 24-hour control CT)
  * Blood pressure, heart rate, oxygen saturation SO2
  * Episodes with severe hypotension with systolic blood pressure <110mmHg
  * Incidence of pneumonia (defined as: any new pulmonary infiltrate on radiographic imaging occurring <48hrs after admission combined with at least one of the subsequent findings: fever >38°C, leukopenia/leucocytosis, purulent secretions with positive cultures)
  * Disturbances in electrolytes, renal function, coagulation (potassium, sodium, chloride, creatinine, INR, pTT, thrombocytes measured on admission before hypothermia and at 24 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Bardutzky, Prof., Principal Investigator — University of Freiburg, Department of Neurology, Germany
Locations (1):
- University of Freiburg, Department of Neurology, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (after anonymization), on which the results of the present study are based, can be made available to scientists upon request (methodologically meaningful evaluation proposal approved by a committee specifically appointed for this evaluation proposal) (6 months to 36 months after publication of the study)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months to 36 months after publication of the study
Access Criteria: upon request of scientists with methodologically meaningful evaluation proposal approved by a committee specifically appointed for this evaluation proposal

REFERENCES:
- See also: Results of the pilot study COTTIS-1 on feasibility and safety — https://svn.bmj.com/content/svnbmj/early/2023/08/22/svn-2023-002420.full.pdf